CLINICAL TRIAL: NCT02436369
Title: The Effect of Yogurt Enriched With Flaxseed on Cardiovascular Risk Factors in Type 2 Diabetic
Brief Title: The Effect of Yogurt Enriched With Flaxseed on Cardiovascular Risk Factors in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Urmia University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: umsu.rec.1393.3
Record Dates: First submitted 2015-04-19; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus
Keywords: diabetic patients; flaxseed; lipid profile; cardiovascular risc factors
MeSH Terms: conditions — Diabetes Mellitus | interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low fat yogurt enriched with flaxseed (Experimental): 200 gr low fat yogurt enriched with 30 gr flaxseed
  Interventions: Dietary Supplement: low fat yogurt enriched with flaxseed
- low fat yogurt (Placebo Comparator): 200 gr low fat yogurt
  Interventions: Dietary Supplement: low fat yogurt

INTERVENTIONS:
Dietary Supplement: low fat yogurt enriched with flaxseed — daily intake of low fat yogurt enriched with flaxseed for 8 weeks
  Arms: low fat yogurt enriched with flaxseed
Dietary Supplement: low fat yogurt — daily intake of low fat yogurt for 8 weeks
  Arms: low fat yogurt

SUMMARY:
The investigators aimed to add flaxseed with high content of n-3 polyunsaturated fatty acids to low fat yogurt to obtain beneficial without adverse effects of it. In this parallel randomized controlled trial the investigators recruited 70 diabetic patients and randomly allocated to control and treatment groups. Participants in treatment group consumed 30 gr flaxseed in 200 gr low fat yogurt, while controls consumed 200 gr just low fat yogurt daily. Lipid profile, fasting blood sugar, glycosylated hemoglobin, systolic and diastolic blood pressure, weight, waist circumference and body mass index were measured at the first and end of the trial.

DETAILED DESCRIPTION:
Nutritionists have concern about consumption of full fat dairy in diabetic patients due to their content of saturated fatty acids. The investigators aimed to add flaxseed with high content of n-3 polyunsaturated fatty acids to low fat yogurt to obtain beneficial without adverse effects of it. In this parallel randomized controlled trial the investigators recruited 70 diabetic patients and randomly allocated to control and treatment groups. Participants in treatment group consumed 30 gr flaxseed in 200 gr low fat yogurt, while controls consumed 200 gr just low fat yogurt daily. Lipid profile, fasting blood sugar, glycosylated hemoglobin, systolic and diastolic blood pressure, weight, waist circumference and body mass index were measured at the first and end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 35 kg/m2 -
* treated with oral hypoglycemic agents (Metformin or Glibenclamide)
* no use of insulin
* fasting blood glucose≥ 126 (but less than 400 mg/dl)or 2 hours blood sugar ≤ 200 mg/dl
* no pregnancy and lactation
* Blood lipids and blood pressure-lowering agents must remained unalteredwithin the last 3 months.

Exclusion Criteria:

* Participants were excluded if they smoked, used alcohol, took dietary supplements containing Omega 3, phytoestrogens, antioxidants and fiber regularly, had been diagnosed with GI disease or renal, liver, cancer , inflammatory disease, had food allergies or intolerances

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in values of FBS at 8 week | 8 weeks
  FBS: Fasting blood sugar
Change from baseline in values of HbA1c at 8 week | 8 weeks
  HbA1C: glycosylated hemoglobin

SECONDARY OUTCOMES:
Change from baseline in values of weight at 8 week | 8 weeks
Change from baseline in values of waist circumference at 8 week | 8 weeks
Change from baseline in values of body mass index at 8 week | 8 weeks
Change from baseline in values of blood pressure at 8 week | 8 weeks
  Blood pressure: systolic blood pressure, diastolic blood pressure
Change from baseline in values of Lipid profile (Total cholesterol, triglyceride, LDL-C, HDL-C) at 8 week | 8 weeks
  Lipid profile:Total cholesterol, triglyceride, LDL-C, HDL-C

REFERENCES:
- [Derived] Hasaniani N, Rahimlou M, Ramezani Ahmadi A, Mehdizadeh Khalifani A, Alizadeh M. The Effect of Flaxseed Enriched Yogurt on the Glycemic Status and Cardiovascular Risk Factors in Patients with Type 2 Diabetes Mellitus: Randomized, Open-labeled, Controlled Study. Clin Nutr Res. 2019 Oct 2;8(4):284-295. doi: 10.7762/cnr.2019.8.4.284. eCollection 2019 Oct. PMID 31720254